CLINICAL TRIAL: NCT03236285
Title: Microvascular and Metabolic Effects of High-intensity Interval Training (HIIT) and Intermittent Fasting (FAST) in Overweight or Obese, Sedentary Women With Cardiometabolic Risk Factors: HIIT-FAST, a Randomized Clinical Trial
Brief Title: Microvascular and Metabolic Effects of High-intensity Interval Exercise Training
Acronym: HIIT-FAST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Facilities for the exercise training program were not available for the study.
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, MD, PhD, National Institute of Cardiology, Laranjeiras, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAAE:69240017.1.0000.5272
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Obesity; Overweight; Physical Activity
Keywords: Obesity; Microcirculation; Endothelial function; Laser speckle imaging; Capillary density
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIIT only (Experimental): Volunteers will be submitted to high-intensity interval training (HIIT) performed in fed state
  Interventions: Behavioral: High-intensity interval exercise training in the fed state
- CT+FAST (Experimental): Volunteers will be submitted to continous training (CT) performed in the fasting state
  Interventions: Behavioral: Continous exercise training in the fasting state
- CT only (Experimental): Volunteers will be submitted to continous training (CT) performed in fed state.
  Interventions: Behavioral: Continous exercise training in the fed state
- HIIT+FAST (Experimental): Volunteers will be submitted to high-intensity interval training (HIIT) performed in the fasting state.
  Interventions: Behavioral: High-intensity interval exercise training in the fasting state

INTERVENTIONS:
Behavioral: High-intensity interval exercise training in the fed state — High-intensity interval exercise training in the fed state
  Arms: HIIT only
Behavioral: Continous exercise training in the fed state — Continous exercise training in the fed state
  Arms: CT only
Behavioral: High-intensity interval exercise training in the fasting state — High-intensity interval exercise training in the fasting state
  Arms: HIIT+FAST
Behavioral: Continous exercise training in the fasting state — Continous exercise training in the fasting state
  Arms: CT+FAST

SUMMARY:
The study investigates the effects of high intensity interval training (HIIT) versus continuous training (CT), combined or not with fasting, on capillary density, microvascular function, cardiometabolic risk markers, functional capacity, and quality of life, in overweight or obese sedentary women with cardiometabolic risk factors. The use of HIIT could promote greater improvements in these parameters than CT. Furthermore, the positive effects of exercise may increase when it is performed in the fasting state, compared to exercise performed in the fed state.

DETAILED DESCRIPTION:
Physical inactivity and increased caloric intake play important roles in the pathophysiology of obesity. Increases of physical activity and modifications of eating behaviors are first-line interventions which, however, are not easily implemented, and lack of time to exercise and difficulties in coping with different diets are common reasons for failure. High-intensity interval training (HIIT) is a "faster" alternative to moderate-intensity continuous training (CT). Conversely, intermittent fasting is also an alternative to more complex diets, as it restricts caloric intake to a specified period of time without major diet composition changes. The combination of HIIT and fasting may therefore provide incremental benefits.

Sedentary women aged ≥ 30 years and ≤50 years, with body mass index ≥25 kg/m2 and cardiometabolic risk factors, will be randomized to HIIT performed in the fasting state, HIIT performed in the fed state, CT in the fasting state or CT in the fed state. Cardiometabolic parameters, anthropometric indices, cardiorespiratory fitness, quality of life and microvascular function (cutaneous capillary density and microvascular reactivity evaluated by laser speckle contrast imaging) will be evaluated before the initiation of the interventions and 4 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age≥ 30 years and ≤50 years
* Premenopausal status
* Body mass index >25 kg/m2
* At least one of the following:

waist circumference ≥80 cm (women); triglycerides ≥150 mg/dl or treatment for this lipid abnormality; High density-lipoprotein cholesterol <50 mg/dl (women), or treatment for this abnormality; fasting plasma glucose ≥100 mg/dl

Exclusion Criteria:

* Any cardiovascular disease, including systemic hypertension
* Diabetes mellitus
* Chronic pulmonary disease
* Any systemic disease or condition that might reduce the adherence or tolerance to exercise or fasting
* Orthopedic or neurologic conditions that might impair exercise training
* Pregnancy or breastfeeding
* Abnormalities elicited at exercise treadmill testing that preclude the initiation of exercise training
* Current engagement in any exercise training protocol

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Capillary density | 6 months
  Number of spontaneously perfused skin capillaries per mm2

SECONDARY OUTCOMES:
Microvascular reactivity assessed by laser speckle contrast imaging | 6 months
  Skin microvascular flow in arbitrary perfusion units

CONTACTS AND LOCATIONS:
Overall Officials: EDUARDO V TIBIRICA, MD, PhD, Principal Investigator — National Innstitute of Cardiology
Locations (1):
- National Institute of Cardiology, Ministry of Health, Brazil, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] De Lorenzo A, Van Bavel D, de Moraes R, Tibirica EV. High-intensity interval training or continuous training, combined or not with fasting, in obese or overweight women with cardiometabolic risk factors: study protocol for a randomised clinical trial. BMJ Open. 2018 Apr 28;8(4):e019304. doi: 10.1136/bmjopen-2017-019304. PMID 29705753